CLINICAL TRIAL: NCT04374812
Title: Consequences, Costs and Cost-effectiveness of Different Workforce Configurations in English Acute Hospitals: a Longitudinal Retrospective Study Using Routinely Collected Data
Brief Title: Workforce Hospital Outcomes (in English Acute Hospitals)
Acronym: WHOs
Status: Completed | Type: Observational
Sponsor: University of Southampton (Other)
Responsible Party: Sponsor
Other Study IDs: NIHR128056; 52957.A1 (Other: Southampton University ERGO II)
Record Dates: First submitted 2020-04-20; First posted 2020-05-05 (Actual); Last update posted 2023-05-31 (Actual); Status verified 2023-05

CONDITIONS: Health Workforce
Keywords: health workforce; outcome measures

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Exposure to registered nurses — Change in outcomes associated with a one hour per patient day increase in exposure to registered nurses
  Other Names: RN staffing level
Other: Exposure to nursing assistants — Change in outcomes associated with a one hour per patient day increase in exposure to nursing assistants
  Other Names: HCA or NA staffing levels

SUMMARY:
Background: The NHS is facing significant challenges in recruiting and retaining staff, particularly registered nurses (RNs). Recruiting unregistered staff is often adopted as a solution to the RN shortage; however recent research found a negative effect of low RN staffing levels on mortality with no evidence that high levels of assistant staff could mitigate the increased risk. Economic modelling suggested that increases in skill mix were potentially cost-effective, but these findings derive from a single NHS hospital Trust with limited cost and outcome data.

Aims and objectives: This project aims to estimate the consequences, costs and cost effectiveness of variation in the size and composition of the staff on hospital wards in England. In order to provide estimates that are more likely to apply across the NHS, this study will include at least four hospitals and consider a wider range of outcomes and sources of costs, including death within 30 days of admission, adverse events such as infections, length of hospital stay, readmissions and rates of staff sickness.

Methods: This retrospective longitudinal observational study will use routinely collected data on ward and shift level nurse staffing, and patient outcomes. Data will be derived from the E-Roster systems, used by hospitals to record all planned and worked shifts. The investigators will consider all rostered direct care staff. These data will be linked to patient data derived from the hospital patient administration system (PAS); and other clinical systems and databases of adverse events (e.g. datix). Relationships between RN and assistant staffing levels and outcomes will be explored using survival models incorporating mixed effects. The investigators will use the results of these analyses to model the costs and consequences of different staffing configurations and to estimate the incremental cost-effectiveness associated with change. Our study will provide evidence to inform staffing levels and skill mix planning in the NHS, highlighting potential cost savings, and offering improved patient safety and reduced adverse staff outcomes.

DETAILED DESCRIPTION:
Note that for this study, "Study start" means the date the first hospital Trust was recruited. "Primary completion" is the date by which the investigators anticipate data analysis for the primary outcomes will be complete. "Study completion" is the data by which investigators anticipate data analysis for secondary outcomes will be complete.

The investigators cannot name the hospital Trusts participating because the investigators do not have their consent and this would breach GDPR.

ELIGIBILITY:
Eligibility criteria for hospitals:

* acute hospital Trust in England
* willingness and ability to provide anonymised patient data and the ability to provide electronic roster data for a minimum period of 1 year prior to the commencement of the study.

Eligibility criteria for patients:

* stayed on at least one acute inpatient ward / admissions unit (including High Dependency Unit and Intensive Care Unit) during the study period.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients staying on inpatient wards in acute hospital Trusts in England
Sampling Method: Non-Probability Sample
Enrollment: 1706388 (Actual)
Dates: Start 2020-09-21 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Patient deaths | 30 days
  Adjusted hazard ratio for death from all causes within 30 days of hospital admission

CONTACTS AND LOCATIONS:
Overall Officials: Peter Griffiths, Principal Investigator — The University of Southampton
Locations (1):
- Hospital Trust A, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Griffiths P, Saville C, Ball J, Culliford D, Jones J, Lambert F, Meredith P, Rubbo B, Turner L, Dall'Ora C. Consequences, costs and cost-effectiveness of workforce configurations in English acute hospitals. Health Soc Care Deliv Res. 2025 Jul;13(25):1-107. doi: 10.3310/ZBAR9152. PMID 40622683
- [Derived] Meredith P, Turner L, Saville C, Griffiths P. Nurse understaffing associated with adverse outcomes for surgical admissions. Br J Surg. 2024 Aug 30;111(9):znae215. doi: 10.1093/bjs/znae215. PMID 39313222
- [Derived] Rubbo B, Saville C, Dall'Ora C, Turner L, Jones J, Ball J, Culliford D, Griffiths P. Staffing levels and hospital mortality in England: a national panel study using routinely collected data. BMJ Open. 2023 May 17;13(5):e066702. doi: 10.1136/bmjopen-2022-066702. PMID 37197808

DOCUMENTS (1):
  • Study Protocol (2022-01-26): https://cdn.clinicaltrials.gov/large-docs/12/NCT04374812/Prot_002.pdf